CLINICAL TRIAL: NCT06201884
Title: Efficacy of Adapted Physical Activity on a Walking Platform in Elderly Patients HOspitalized for Cancer Surgery
Acronym: APPAHOCA-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-A01292-43
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Oncology; Elderly Patients; Surgery
Keywords: Adapted physical activity; walking platform
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adapted physical activity (Experimental): Adapted physical activity on a walking platform
  Interventions: Device: Early rehabilitation through Adapted Physical Activity

INTERVENTIONS:
Device: Early rehabilitation through Adapted Physical Activity — From the day after surgery, 1 to 2 walking sessions with walking platform, lasting 6 to 30 minutes (min-max), will be proposed daily until the day of discharge.

SUMMARY:
The aim of this study was to evaluate the efficacy of daily use of a walking platform to improve recovery of preoperative walking speed at hospital discharge following oncological surgery in patients aged 65 or older.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 65 or over
* Candidate for scheduled major oncological surgery and/or surgery with high morbidity
* Patient able to walk for 10 minutes on the walking platform at the time of the test
* Patient affiliated to a social security system
* Signature of informed consent prior to any specific study-related procedure

Exclusion Criteria:

* Patient with severe undernutrition (BMI<18, and/or weight loss >15% in 6 months or >10% in 1 month)
* Emergency surgery
* Physical contraindications preventing use of the platform
* Simultaneous participation in another clinical study that could compromise the conduct of this study
* Patients deprived of their liberty, under guardianship or subject to a legal protection measure, or unable to express their consent.
* Patient unable to undergo trial follow-up for geographical, social or psychopathological reasons.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of daily use of a walking platform to improve recovery of preoperative walking speed at hospital discharge following oncological surgery in patients aged 65 or older. | at hospital discharge (approximately 15 to 30 days after surgery)
  Proportion of patients having recovered their preoperative walking speed at hospital discharge

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Francois Baclesse, Caen
  - CHU CAEN, Caen

IPD SHARING:
Plan to Share IPD: Undecided